CLINICAL TRIAL: NCT01115257
Title: Severe Proliferative Diabetic Retinopathy Treated With Vitrectomy or Panretinal Photocoagulation: a Prospective Comparative Study
Brief Title: Severe Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Prof. Teresio Avitabile, 1Department of Medicine and Surgery, Section of Ophthalmology, Santa Marta Hospital, University of Catania, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0016258
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2006-10

CONDITIONS: Diabetic Retinopathy
Keywords: severe proliferative diabetic retinopathy; vitrectomy; panretinalphotocoagulation
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Other): 90 eyes of 90 patients, with severe PDR, some with tractional retinal detachment (TRD) not involving the macula were included in the study and treated with vitrectomy
  Interventions: Procedure: vitrectomy
- panretinalphotocoagulation (group 2) (Other): 90 eyes of 90 patients, with severe PDR, some with tractional retinal detachment (TRD) not involving the macula were included in the study and treated with panretinalphotocoagulation
  Interventions: Procedure: panretinalphotocoagulation

INTERVENTIONS:
Procedure: vitrectomy — The surgical technique (Group 1) included vitrectomy, with a combination of delamination and segmentation of gliotic tractional membranes using bimanual technique. Silicone oil tamponade was used in eyes with long-standing tractional retinal detachment, as deemed necessary by the surgeon, or in eyes in which a retinal break occurred during the vitrectomy.
  Arms: group 1
Procedure: panretinalphotocoagulation — Panretinal photocoagulation was completed according to guidelines summarized in ETDRS with extensive full subconfluent panretinal photocoagulation.
  Arms: panretinalphotocoagulation (group 2)

SUMMARY:
The purpose of this study is to examine and compare, prospectively, best corrected visual acuity (BCVA) outcomes and complications of a cohort of patients with Proliferative Diabetic Retinopathy and Tractional Retinal Detachment not involving macula undergoing pars plana vitrectomy (PPV) or conventional management (panretinal photocoagulation).

DETAILED DESCRIPTION:
The utility and practice of Panretinalphotocoagualtion (PRP) in patients with high-risk Proliferative Diabetic Retinopathy (PDR) have not changed since the ETDRS reported guidelines in 1987. A meta-analysis of the DRS and ETDRS two large U.S. RCT of laser therapy for PDR confirmed the effectiveness of PRP (Level I evidence). Both trials had large sample sizes, excellent compliance and adequate follow-up. These studies established that PRP reduces the risk of severe visual loss in patients with high-risk PDR by 50% to 60%20.

With the arrival of the vitrectomy, this surgery was often used to treat eyes with severe complications from PDR. The most common indications for vitrectomy were nonclearing vitreous hemorrhage, Tractional Retinal Detachment(TRD) with macular involvement, and combined traction and rhegmatogenous retinal detachment. With the addition of new indications to the known indications vitrectomy has been performed in earlier stages(severe PDR). A large number of case series reports have assessed the effect of pars plana vitrectomy on diabetic TRD with or without macular detachment but the level of evidence was low and they included patients not homogeneous. These studies have generally shown benefit, with improved vision seen in many patients (ranging from 22% to 65%) but they have also indicated a high rate of operative and postoperative complications. These numerous intra and post-operative complications could lead to satisfying anatomical results but poor vision.The purpose of this study is to examine and compare, prospectively, best corrected visual acuity (BCVA) outcomes and complications of a cohort of patients with Proliferative Diabetic Retinopathy and Tractional Retinal Detachment not involving macula undergoing pars plana vitrectomy (PPV) or conventional management (panretinal photocoagulation)

ELIGIBILITY:
Inclusion Criteria:

* Eyes with advanced Proliferative diabetic retinopathy some with TRD not involving the macula. The definition of severe PDR included eyes with extensive, active neovascular and fibrovascular proliferation graded using Modified Airlie House Classification

Exclusion Criteria:

* Eyes with fibrovascular tractional detachment involving the macula were excluded. Eyes with a combined tractional and rhegmatogenous retinal detachment and eyes with a history of uveitis or trauma, with previous vitrectomy and neovascular glaucoma were also excluded.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2001-10; Primary Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresio Avitabile, Professor, Study Chair — universita studi di Catania
Locations (1):
- 1Department of Medicine and Surgery, Section of Ophthalmology, Santa Marta Hospital, University of Catania, Italy, Catania, Italy, Italy

REFERENCES:
- [Derived] Avitabile T, Bonfiglio V, Castiglione F, Castaing M, Contarino F, Mistretta A. Severe proliferative diabetic retinopathy treated with vitrectomy or panretinal photocoagulation: a monocenter randomized controlled clinical trial. Can J Ophthalmol. 2011 Aug;46(4):345-51. doi: 10.1016/j.jcjo.2011.06.012. Epub 2011 Jul 7. PMID 21816255